CLINICAL TRIAL: NCT05755126
Title: The Comparative Efficacy of Iatrosedation and Music Therapy as Techniques to Attenuate Dental Anxiety in Patients Undergoing Dental Crown Preparation
Brief Title: Efficacy of Iatrosedation and Music Therapy to Attenuate Dental Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Altamash Institute of Dental Medicine (Other)
Responsible Party: Principal Investigator, Abhishek Lal, Principal Investigator, Altamash Institute of Dental Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Iatrosedation vs Music
Record Dates: First submitted 2023-02-14; First posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: Dental Anxiety

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Iatrosedation (Experimental)
  Interventions: Behavioral: Iatrosedation
- Musical Therapy (Experimental)
  Interventions: Behavioral: Musical Therapy
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Iatrosedation — Alleviating the anxiety of patients by iatrosedative interview and clinical encounter
  Arms: Iatrosedation
Behavioral: Musical Therapy — Patients were provided with headphones and a playlist to listen to the music of their choice for 10 minutes
  Arms: Musical Therapy

SUMMARY:
Dental anxiety is a common problem encountered in the dental clinics that affect both patients and dentists. Adequate management of the dental anxiety is critical for optimal treatment outcomes of the patient. In this clinical trial, a total of sixty patients were randomly assigned to three groups as follows: Group 1, Iatrosedation, Group 2, Music Therapy, and Group 3, Control. Patients in all of the three groups underwent dental crown preparation. . To measure the anxiety levels of the patients, heart rate was measured using a pulse oximeter, and verbal rating scale scores were assessed

DETAILED DESCRIPTION:
Dental anxiety is a common problem encountered in the dental clinics that affect both patients and dentists. Adequate management of the dental anxiety is critical for optimal treatment outcomes of the patient.

This study aims to assess the efficacy of different anxiety reduction techniques (Iatrosedation and music therapy) in adult patients for dental crown preparations.

In this clinical trial, a total of sixty patients were randomly assigned to three groups as follows: Group 1, Iatrosedation, Group 2, Music Therapy, and Group 3, Control. Patients in all of the three groups underwent dental crown preparation. To measure the anxiety levels of the patients, heart rate was measured using a pulse oximeter, and verbal rating scale scores were assessed. One-way ANOVA, Post hoc, and Spearman's correlation was used to compare the mean values of the three groups.

ELIGIBILITY:
Inclusion Criteria:

* patients who were above 18 years of age
* no systemic diseases
* no previous dental treatment experience
* showed willingness to participate

Exclusion Criteria:

* patients below the age of 18 years
* medically compromised
* previous history of dental treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Dental Anxiety | 6 months
  Heart rate was measured using a pulse oximeter
Dental Anxiety | 6 months
  Using verbal rating scale scores

CONTACTS AND LOCATIONS:
Locations (1):
- Altamash Institute of Dental Medicine, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided